CLINICAL TRIAL: NCT00791830
Title: Saving Residual Renal Function Among Haemodialysis Patients Receiving Irbesartan - a Double Blind Randomised Study
Brief Title: Saving Residual Renal Function Among Haemodialysis Patients Receiving Irbesartan
Acronym: SAFIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT no: 2008-001267-11
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Residual renal function; Haemodialysis; Applanation tonometry; Cardiac output; Quality of life; Angiotensin II Type 1 Receptor Blockers
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irbesartan (Active Comparator)
  Interventions: Drug: Irbesartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching irbesartan 150 mg

INTERVENTIONS:
Drug: Irbesartan — Tablets, 300 mg * 1 daily, 1 year
  Other Names: Aprovel; Karvea; Avapro; CAS no: 138402-11-6; ATC code: C09CA04; PubChem: 3749; Drugbank: APRD00413
  Arms: Irbesartan
Drug: Placebo matching irbesartan 150 mg — Tablets, 300 mg * 1 daily, 1 year
  Arms: Placebo

SUMMARY:
Angiotensin II receptor blockers (ARB) are known to preserve kidney function among patients with kidney diseases and reduced renal function, but not among haemodialysis patients.

Haemodialysis patients often lose residual renal function after initiating dialysis leading to worsened quality of life, increased morbidity and mortality.

In this study an ARB is investigated in a double blind, randomised, parallel group, placebo controlled manner to see, if this ARB can save residual renal function among haemodialysis patients. Potential cardiovascular benefits of the treatment are also addressed.

DETAILED DESCRIPTION:
Haemodialysis patients often lose residual renal function rather quickly after initiation of dialysis - average loss is 30 % per year. Loss of residual kidney function leads to deteriorating quality of life, more morbidity and a higher mortality. Many causes to this has been identified, but no one has - to my knowledge - addressed saving of residual renal function among haemodialysis patients so far.

Hypothesis: Irbesartan can reduce loss of residual kidney function among haemodialysis patients and left ventricular hypertrophy and arterial stiffness is less pronounced after 1 year of treatment.

Methods: 80 patients are randomised to receive either irbesartan, an angiotensin II receptor blocker (ARB), or placebo for 1 year. Residual renal function will be estimated before and one-two weeks after initiating project medicine, in order to estimate the acute effect of ARB on residual renal function in this study population. Thereafter, glomerular filtration rate (GFR) and urine volume will be determined after 3, 6, 9 and 12 months giving a regression line for each patient. 8 dialysis units will be recruiting patients.

Investigations:

* creatinine-urea-clearance by 24h urine collection
* applanation tonometry
* cardiac output
* echocardiography
* QoL questionnaire
* endocrinological and cardiovascular markers in blood and urine

Perspectives: It is well-known that ceased urine production has a tremendous negative effect on the quality of life of haemodialysis patients. Lately it was shown that residual renal function has greater impact than dialysis dose on morbidity as well as mortality. Among peritoneal dialysis patients in Asia an angiotensin-converting enzyme inhibitors (ACEI) or an ARB saved residual renal function, but preservation of renal function has not been addressed in haemodialysis patients, and ACEI or ARB are only prescribed to roughly 15 % of these.

If this study confirms our hypothesis the growing population of haemodialysis patients should be offered irbesartan.

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis patient
* Haemodialysis treatment for maximum 12 months
* > 18 years old
* informed consent
* urine volume > 300 ml / 24 hours
* contraception if fertile woman

Exclusion Criteria:

* Systolic blood pressure < 110 mm Hg
* Able to comprehend the aims of the project and follow instructions
* Allergy to irbesartan/ACE-inhibitors/ARBs
* Myocardial infarction or unstable angina pectoris during the last 3 months
* Ejection fraction < 30 %
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Decrease in loss of residual kidney function. | 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Cardio-vascular outcome assessed by applanation tonometry, echocardiography, Transonic measurements of cardiac output and markers in blood. | 1 year
Progression to anuria | 3, 6, 9 and 12 months
Quality of life assessed by a questionnaire: Kidney Disease Quality Of Life - Short Form (KDQOL-SF) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bente Jespersen, MD, DrMedSc, Study Chair — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Erik Sloth, MD, DrMedSc, Study Chair — Department of Anaesthesiology and Intensive Care, Aarhus University Hospital, Skejby, Denmark; Jens Kristian D Jensen, MD, PhD, Study Chair — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Krista D Kjærgaard, MD, PhD, Study Director — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Christian D Peters, MD, Study Chair — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Charlotte Strandhave, MD, Principal Investigator — Department of Nephrology, Aalborg University Hospital, Denmark; Ida N Tietze, MD, PhD, Principal Investigator — Department of Internal Medicine, Region Hospital Viborg, Denmark; Marija K Novosel, MD, Principal Investigator — Department of Internal Medicine, Region Hospital Fredericia, Denmark
Locations (6):
- Denmark (6):
  - Department of Nephrology, Aarhus University, Aalborg, Aalborg
  - Department of Nephrology, Aarhus University Hospital, Skejby, Aarhus N
  - Department of Medicine, Fredericia Hospital, Fredericia
  - Haemodialysis unit, Horsens Hospital, Horsens
  - Hemodialysis Unit, Randers Hospital, Randers
  - Department of Medicine M, Viborg Hospital, Viborg

REFERENCES:
- [Derived] Peters CD, Kjaergaard KD, Christensen KL, Bibby BM, Jespersen B, Jensen JD. High-sensitivity Troponin T in hemodialysis patients: a randomized placebo-controlled sub-study investigating angiotensin-II-blockade, variation over time and associations with clinical outcome. BMC Nephrol. 2020 Oct 28;21(1):452. doi: 10.1186/s12882-020-02103-1. PMID 33115436
- [Derived] Peters CD, Kjaergaard KD, Jensen JD, Christensen KL, Strandhave C, Tietze IN, Novosel MK, Bibby BM, Jespersen B. Short and Long-Term Effects of the Angiotensin II Receptor Blocker Irbesartan on Intradialytic Central Hemodynamics: A Randomized Double-Blind Placebo-Controlled One-Year Intervention Trial (the SAFIR Study). PLoS One. 2015 Jun 1;10(6):e0126882. doi: 10.1371/journal.pone.0126882. eCollection 2015. PMID 26030651
- [Derived] Peters CD, Kjaergaard KD, Jespersen B, Christensen KL, Jensen JD. Renal and cardiovascular effects of irbesartan in dialysis patients--a randomized controlled trial protocol (SAFIR study). Dan Med J. 2013 Apr;60(4):A4602. PMID 23651713